CLINICAL TRIAL: NCT04984460
Title: A Multicenter Clinical Study on Liquid-based Morphological Detection of Fungi
Brief Title: Morphological Detection of Liquid-based Thin-layer Film-making Fungi for Fungal Vaginitis in Multiple Hospitals
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Affiliated Hospital of Nantong University (Other)
Responsible Party: Principal Investigator, Yuquan Zhang, Director of Obstetrics and Gynaecology, Affiliated Hospital of Nantong University
Other Study IDs: AHNantongU_YEZH_NTFS_V1.0
Record Dates: First submitted 2021-07-22; First posted 2021-07-30 (Actual); Last update posted 2021-07-30 (Actual); Status verified 2021-07

CONDITIONS: Vaginitis
Keywords: Fluorescence morphological; liquid-based thin-layer film-making; Fungal vaginitis
MeSH Terms: conditions — Vaginitis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- life-style counseling: A sample of one or more of the following characteristics. Symptoms: vulva pruritus, burning pain, but also accompanied by pain in urine and sexual pain and other symptoms; Leucorrhea increased.
  Physical signs: Vulva flushing, edema, visible scratches or chaps, white membrane attached to the inner side of the labia minora and the vaginal mucosa, more white bean residue like secretions can be seen in the vagina, which can be curd.
  Interventions: Diagnostic Test: Fluorescence morphological detection of liquid-based thin-layer film-making fungi

INTERVENTIONS:
Diagnostic Test: Fluorescence morphological detection of liquid-based thin-layer film-making fungi — Samples from outpatient or inpatient clinics to be tested for fungal vaginitis. A sample of one or more of the following characteristics. Symptoms: vulva pruritus, burning pain, but also accompanied by pain in urine and sexual pain and other symptoms; Leucorrhea increased.
  Physical signs: Vulva flushing, edema, visible scratches or chaps, white membrane attached to the inner side of the labia minora and the vaginal mucosa, more white bean residue like secretions can be seen in the vagina, which can be curd.
  Samples are human vaginal secretions. Each sample should be the amount on one swab.
  The sample is not in menstrual period. The sample subjects did not have vaginal irrigation, medication or sexual intercourse within 3 days.

SUMMARY:
The purpose of this study is to compare the results of different detection methods for non-gestational fungal vaginitis (VVC), and to evaluate the significance of different fungal states in the results for diagnosis and treatment.

DETAILED DESCRIPTION:
The study was divided into two phases: in the first phase, the vaginal secretions of 1000 enrolled patients with fungal vaginitis were detected with 3/4 different methods, and the sensitivity, specificity and consistency of these methods were compared; In the second stage, 1000 patients from the first stage were selected to meet the follow-up stage and divided into two groups. The test of Follow-up fungal culture and fluorescence morphological detection of liquid-based thin-layer film-making fungi were performed periodically. At last, the applicant will analyze the data, write the paper and publish the article.

ELIGIBILITY:
Inclusion Criteria:

* 1. Samples from outpatient or inpatient clinics to be tested for fungal vaginitis.
* 2. A sample of one or more of the following characteristics. 2.1 Symptoms: vulva pruritus, burning pain, but also accompanied by pain in urine and sexual pain and other symptoms; Leucorrhea increased.

2.2 Physical signs: Vulva flushing, edema, visible scratches or chaps, white membrane attached to the inner side of the labia minora and the vaginal mucosa, more white bean residue like secretions can be seen in the vagina, which can be curd.

* 3. The samples are vaginal secretions from the female body. Each sample should be the amount on one swab.
* 4. The sample is not in menstrual period.
* 5. The sample subjects did not have vaginal irrigation, medication or sexual intercourse within 3 days.

Exclusion Criteria:

* 1. Cases with incomplete specimen collection;
* 2. Mixed vaginitis cases;
* 3. Abscission cases with incomplete follow-up.

Ages: 14 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Fungal vaginitis is a disease that only women get.
Study Population: Female patients with suspected fungal vaginitis.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2021-07-09 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-04-01 (Estimated)

PRIMARY OUTCOMES:
Comparing the positive detection rate of 3/4 different detection methods in the first phase. | From Aug. 1st to Dec. 31st, 2021
  The positive coincidence rate (sensitivity), negative coincidence rate (specificity) and total coincidence rate (consistency) was compared, according to the P<0.05 was used to determine whether it was statistically significant.
Calculating the proportion of the number of fungi in three different states in the map results of three/four detection methods. | From Aug. 1st, 2021 to Jan. 31st, 2022
  Counting The number and proportion of mycelia, spores and blastospores, especially the percentage of cases of single spore (+) in all cases of fungus (+).
Counting the positive numbers of 4 or 6 liquid-based thin-layer fungal fluorescence morphological tests and fungal culture in the Stage 2_follow-up stage. | From Mar. 1, 2022 to Dec. 31st, 2022
  the positive coincidence rate (sensitivity), negative coincidence rate (specificity) of 4 or 6 liquid-based thin-layer fungal fluorescence morphological tests

CONTACTS AND LOCATIONS:
Overall Officials: Yuquan Zhang, Doctor, Principal Investigator — Affiliated Hospital of Nantong University
Locations (10):
- China (10):
  - The First Affiliated Hospital of Ustc, Hefei, Anhui
  - Zhongshan City People's Hospital, Zhongshan, Guangdong
  - The Second Affiliated Hospital of Nantong University, Nantong, Jiangsu
  - Affiliated Hospital of Nantong University, Nantong, Jiangsu
  - Affiliated Nantong Hospital Of Shanghai University, Nantong, Jiangsu
  - Nantong Maternal and Child Health Hospital, Nantong, Jiangsu
  - Children's Hospital of Fudan University Qidong Branch, Qidong, Jiangsu
  - Jiujiang Maternal and Child Health Hospital, Jiujiang, Jiangxi
  - Jiangxi Maternal and Child Health Hospital, Nanchang, Jiangxi
  - Changning District Maternal and Child Health Care Hospital, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No
Not planning sharing at present.